CLINICAL TRIAL: NCT00690378
Title: Prospective, Multicenter, Investigator-blinded, Randomized, Comparative Study Estimate Safety, Tolerability, Efficacy of NXL104/Ceftazidime vs. Comparator Followed Appropriate Oral Therapy Treatment Complicated UTI Hosp Adults
Brief Title: Comparative Study of NXL104/Ceftazidime Versus Comparator in Adults With Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NXL104/2001; C3591013 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-04 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-03

CONDITIONS: Complicated Urinary Tract Infection
MeSH Terms: interventions — avibactam; Ceftazidime; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): NXL/104 ceftazidime
  Interventions: Drug: NXL104/ceftazidime
- 2 (Active Comparator): comparator 4 x daily
  Interventions: Drug: Imipenem/Cilastatin

INTERVENTIONS:
Drug: NXL104/ceftazidime — 125mg/500mg TID
  Arms: 1
Drug: Imipenem/Cilastatin — 4 x daily
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether NXL104 plus ceftazidime is effective in the treatment of complicated urinary tract infections as compared to a comparator group.

ELIGIBILITY:
Inclusion Criteria:

* Acute pyelonephritis or other complicated urinary tract infection due to gram negative pathogens

Exclusion Criteria:

* ileal loops or vesicoureteral reflux
* complete obstruction of any portion of urinary tract, perinephric or intrarenal abscess.
* fungal urinary tract infection
* permanent indirect catheter or nephrostomy unless removed within 48 hours of study entry
* history hypersensitivity to study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Carole A Sable, MD, Study Director — Novexel Inc
Locations (59):
- United States (42):
  - Alabama Research Center, Birmingham, Alabama
  - Southeast Alabama Medical Center, Dothan, Alabama
  - Providence Hospital, Mobile, Alabama
  - Arizona Pulmonary Specialists LTD, Phoenix, Arizona
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Synergy Clinical Research Center, Escondido, California
  - Novellus Research Sites, Fountain Valley, California
  - Novellus Research Sites, Long Beach, California
  - Modesto Clinical Research, Modesto, California
  - Tri City Medical Center, Oceanside, California
  - EStudy Site, San Jose, California
  - Olive View UCLA Medical Center, Sylmar, California
  - Christiana Care Health Services, Newark, Delaware
  - Century Clinical Research, Inc, Daytona Beach, Florida
  - University of Florida, Jacksonville, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - Louisiana State University Health Services Ctr Shreveport, Shreveport, Louisiana
  - R. Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - North Memorial Medical Center, Minneapolis, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - St. James Healthcare, Butte, Montana
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University Hospital UMDNJ, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Brookdale University Hospital, Brooklyn, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Staten Island University Hospital, Staten Island, New York
  - Mission Hospital, Asheville, North Carolina
  - Clinical Trials of America Inc., Winston-Salem, North Carolina
  - Summa Health System Hospitals, Akron, Ohio
  - Remington-Davis, Columbus, Ohio
  - Regional Infectious Disease-Infusion Center, Lima, Ohio
  - St Vincent's Mercy Medical Center, Toledo, Ohio
  - Thomas Jefferson Univ Hospital, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Harris Methodist, Azle, Texas
  - University of Texas MD Anderson, Houston, Texas
  - Sentara Norfold General Hospital, Norfolk, Virginia
- Jordan (4):
  - Al-Essra hospital, Amman
  - Al-Islami Hospital, Amman
  - Jordan University Hospital, Amman
  - King Abdullah University Hospital, Irbid
- Lebanon (13):
  - Clinique due Levant Hospital, Beirut
  - Dr. Rizk Clinic, Beirut
  - Makassed General Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Sahel General Hospital, Beirut
  - Notre Dame Des Secours Hospital, Byblos
  - Ain Wazein Hospital, Chouf
  - St. Joseph Hospital, Ed Daoura
  - Mount Lebanon Hospital, Hazmiyeh
  - Nabatyeh Governmental Hospital, Nabatyeh
  - Hammoud Hospital University Medical Center, Saida
  - Labib Medical Center, Saida
  - Saida Governmental Hospital, Saida

REFERENCES:
- [Derived] Vazquez JA, Gonzalez Patzan LD, Stricklin D, Duttaroy DD, Kreidly Z, Lipka J, Sable C. Efficacy and safety of ceftazidime-avibactam versus imipenem-cilastatin in the treatment of complicated urinary tract infections, including acute pyelonephritis, in hospitalized adults: results of a prospective, investigator-blinded, randomized study. Curr Med Res Opin. 2012 Dec;28(12):1921-31. doi: 10.1185/03007995.2012.748653. Epub 2012 Nov 21. PMID 23145859

RESULTS

PARTICIPANT FLOW:
Groups:
- NXL104/CAZ: NXL104 125mg/Ceftazidime 500mg TID
- Imipenem Cilastatin: Imipenem cilastatin 500mg 4xdaily
Period: Overall Study
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Started | 69 (Randomized) | 68 (Randomized)
Treated | 68 | 67
Completed | 49 (Up to Late follow up (LFU) visit) | 54 (Up to LFU visit)
Not Completed | 20 | 14
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Did not meet inc/exc criteria | 13 | 11
Not completed — Social problem | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | NXL104/CAZ | Imipenem Cilastatin | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (18.24) | 49.9 (18.44) | 48.15 (18.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Microbiological Outcome at the Test of Cure (TOC) Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 19 | 25

2. Secondary Outcome: Clinical Outcome in Clinically Evaluable (CE) Patients at the End of Intravenous (IV) Therapy Visit
Description: Cure: all or most pre-therapy signs and symptoms of the index infection had resolved and no additional antibiotic was required
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 28 | 36
Participants | 28 | 36

3. Secondary Outcome: Clinical Outcome in CE Patients at the TOC Visit
Description: as for outcome 2
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 28 | 36
Participants | 24 | 29

4. Secondary Outcome: Clinical Outcome in CE Patients at the Late Follow-up (LFU) Visit
Description: Cure: all or most pre-therapy signs and symptoms of the index infection showed no evidence of resurgence and no additional antibiotic was required
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 36
Participants | 20 | 24

5. Secondary Outcome: Microbiological Outcome in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 25 | 34

6. Secondary Outcome: Microbiological Outcome in ME Patients at the LFU Visit
Description: Sustained eradication: a uropathogen found at entry at >10^5 CFU/mL remained <10^4 CFU/mL
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 26 | 30
Participants | 15 | 18

7. Secondary Outcome: Microbiological Outcome for the Urine Pathogen C. Koseri in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 1 | 0

8. Secondary Outcome: Microbiological Outcome for the Urine Pathogen E. Cloacae in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 1

9. Secondary Outcome: Microbiological Outcome for the Urine Pathogen E. Coli in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 24 | 32
Participants | 24 | 32

10. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Mirabilis in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 1

11. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Aeruginosa in ME Patients at the End of IV Therapy Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: End of IV therapy (4 to 14 days)
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 1 | 0

12. Secondary Outcome: Microbiological Outcome for the Urine Pathogen C. Koseri in ME Patients at the TOC Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 1 | 0

13. Secondary Outcome: Microbiological Outcome for the Urine Pathogen E. Cloacae in ME Patients at the TOC Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 1

14. Secondary Outcome: Microbiological Outcome for the Urine Pathogen E. Coli in ME Patients at the TOC Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 25 | 33
Participants | 19 | 23

15. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Mirabilis in ME Patients at the TOC Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 1

16. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Aeruginosa in ME Patients at the TOC Visit
Description: Eradication: a uropathogen found at entry at >10^5 CFU/mL was reduced to <10^4 CFU/mL
Time Frame: 5 to 9 days post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 0

17. Secondary Outcome: Microbiological Outcome for the Urine Pathogen C. Koseri in ME Patients at the LFU Visit
Description: Sustained eradication: a uropathogen found at entry at >10^5 CFU/mL remained <10^4 CFU/mL
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 1 | 0

18. Secondary Outcome: Microbiological Outcome for the Urine Pathogen E. Coli in ME Patients at the LFU Visit
Description: Sustained eradication: a uropathogen found at entry at >10^5 CFU/mL remained <10^4 CFU/mL
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 24 | 29
Participants | 15 | 17

19. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Mirabilis in ME Patients at the LFU Visit
Description: Sustained eradication: a uropathogen found at entry at >10^5 CFU/mL remained <10^4 CFU/mL
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 1

20. Secondary Outcome: Microbiological Outcome for the Urine Pathogen P. Aeruginosa in ME Patients at the LFU Visit
Description: Sustained eradication: a uropathogen found at entry at >10^5 CFU/mL remained <10^4 CFU/mL
Time Frame: 4 to 6 weeks post-therapy
Measure: Number; unit: Participants
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Number analyzed (Participants) | 27 | 35
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 19 days
Arm/Group | NXL104/CAZ | Imipenem Cilastatin
Serious Adverse Events (participants affected / at risk) | 6/68 | 2/67
Other Adverse Events (participants affected / at risk) | 30/68 | 33/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NXL104/CAZ (N=68) | Imipenem Cilastatin (N=67)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NXL104/CAZ (N=68) | Imipenem Cilastatin (N=67)
Constipation (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 7
Abdominal Distension (Gastrointestinal disorders) | 0 | 5
Abdominal Pain (Gastrointestinal disorders) | 5 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 1
Infusion Site Reaction (General disorders) | 2 | 10
Injection Site Reaction (General disorders) | 3 | 6
Chest Pain (General disorders) | 4 | 3
Alanine Aminotransferase Increased (General disorders) | 2 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 13 | 21
Dizziness (Nervous system disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 7 | 5
Insomnia (Psychiatric disorders) | 4 | 4
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.